CLINICAL TRIAL: NCT04507035
Title: Study on the Treatment of Refractory and Locally Advanced Head and Neck Malignant Tumor With Anlotinib Hydrochloride Capsules Combined With Chemoradiotherapy
Brief Title: Treating Locally Advanced Head and Neck Malignant Tumor With Anlotinib and Chemoradiotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Clinical professor. Zhen-Wei Peng, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: head and neck cancer 007
Record Dates: First submitted 2020-07-17; First posted 2020-08-10 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Anlotinib treatment plus chemoradiotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib group (Experimental): After 2 cycles of anlotinib treatment, we evaluate the therapeutic effect of tumor treatment: If it achieve downgrading and is operable, surgical treatment will be performed; if it is still inoperable and could accept radiotherapy, radiotherapy and chemotherapy will be combined with oral chemotherapy of anlotinib until the end of radiotherapy. Efficiency and side effects will be evaluated within 3 months after therapy. Finally, the survival is in follow-up.
  Interventions: Drug: Anlotinib hydrochloride capsules

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsules — Using anlotinib of 2 cycles as the first-line therapy.
  Other Names: Fukewei, YBH00802018

SUMMARY:
Head and neck tumors include well-differentiated squamous cell carcinoma, adenocarcinoma, adenoid cystic carcinoma, small cell carcinoma, sarcoma, olfactory blastoma, and mucoepidermoid carcinoma, which are highly invasive and have a high rate of recurrence and metastasis. For tumors that cannot be radically removed at the local advanced stage, even after traditional comprehensive treatment, survival is still very low. Therefore, we need to explore new treatment methods to achieve tumor degeneration and increase the surgical resection rate or control local lesions to improve the survival rate of tumors. According to previous research reports and clinical exploration, anlotinib has evidence support for the treatment of locally advanced head and neck tumors. With a considerable effect in the early stage, we tried to initially observe the clinical treatment efficiency, toxic and side effects, progression-free survival time, overall survival time and quality of life of anlotinib in the treatment of patients with refractory head and neck carcinoma. Provide patients with a more optimal treatment plan and improve survival.

DETAILED DESCRIPTION:
We will prospectively collect 30 patients who receive anlotinib combined with chemoradiotherapy. Data will be stored in a private database. The process of data collection will be supervised and regular data examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years;
* Performance status (PS) score ≤ 1 points;
* The expected survival period is more than 3 months;
* Highly differentiated squamous cell carcinoma or non-squamous cell carcinoma of the head and neck diagnosed by pathology and/or cytology, including sarcoma, adenoid cystic carcinoma, olfactory blastoma, mucoepidermoid carcinoma, etc.; those whose primary tumor cannot be cured by surgery;
* With measurable lesions: According to the evaluation criteria for the efficacy of solid tumors (Response Evaluation Criteria In Solid Tumors 1.1), the patient has at least one measurable lesion. The measurable lesion should not have received local treatment such as radiotherapy (target lesion located in the previous radiotherapy area, if it is confirmed that significant progress has occurred , And comply with evaluation standard, can also be used as target lesions);
* No previous anti-tumor therapy, including anti-angiogenesis therapy, such as pazopanib, sunitinib, sorafenib, regorafenib, etc.;
* Sufficient liver function: total bilirubin ≤ upper limit of normal value (ULN); glutamic oxalacetic transaminase (AST) and glutamic-pyruvic transaminase (ALT) ≤ 2 times upper limit of normal value (ULN); alkaline phosphatase ≤ 5 times upper limit of normal value (ULN);
* Adequate renal function: creatinine clearance rate ≥80 mL/min;
* Adequate blood function: absolute neutrophil count (ANC) ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥9g/dL;
* No serious heart, lung and other important organ dysfunction;
* Women of childbearing age must have taken reliable contraceptive measures; pregnancy tests (serum or urine) are negative within 7 days before enrollment, and must be non-lactating patients; and are willing to adopt appropriate during the test and within 6 months after the last treatment Methods of contraception. For men, it is necessary to agree to use appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last dose;
* The subjects voluntarily joined the study and signed an informed consent form with good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Can undergo radical surgery or cannot tolerate anti-tumor treatment;
* Women who are pregnant or breastfeeding, have fertility but are unwilling or unable to take effective contraceptive measures;
* People with high blood pressure who cannot be well controlled by antihypertensive drugs (systolic blood pressure> 150 mmHg, diastolic blood pressure> 100 mmHg);
* Patients with clinically significant cardiovascular disease within 6 months before enrollment, including uncontrolled hypertension, myocardial infarction, or unstable angina; New York Heart Association (NYHA) congestive heart failure of grade II or higher, severe Of arrhythmia requiring treatment (including QT interval ≥440 ms), or cardiac ejection fraction <50%, peripheral vascular disease of grade II or higher;
* Abnormal blood coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or activated partial thromboplastin time (APTT) >1.5 ULN), have bleeding tendency or are undergoing thrombolysis or anticoagulation treatment;
* There was obvious hemoptysis blood 2 months before enrollment, or the daily hemoptysis amount was 2.5ml or more;
* Significant clinically significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline occult blood ++ and above, or suffering from vasculitis within 3 months before enrollment; Known hereditary or acquired bleeding and thrombotic tendency;
* Arterial/venous thromboembolic events within 12 months before enrollment;
* Have undergone major surgery within 4 weeks of enrollment or accompanied by severe, non-healing wounds, ulcers or fractures;
* There are obvious factors that affect the absorption of oral drugs;
* Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred 6 months before enrollment;
* Urinary routines suggest that urine protein is ≥++, and that the amount of urine protein in 24 hours is ≥1.0g;
* Serous cavity fluid accumulation with clinical symptoms and requiring symptomatic treatment;
* Active infections require antimicrobial treatment;
* Have a history of central nervous system diseases, including primary brain tumors, seizures without standard medication, any brain metastases or have cerebrovascular accidents (CVA, stroke), transient ischemic attack (TIA), or 6 A history of subarachnoid hemorrhage within the month;
* Participated in clinical trials of other drugs 4 weeks before enrollment;
* Other malignant tumors in the past or at the same time (except for malignant tumors that have been cured and survived for more than 5 years without cancer, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma, etc.);
* Those who have received VEGFR inhibitors, such as pazopanib, sunitinib, sorafenib, regorafenib, etc.;
* Those who are known to have a history of psychotropic substance abuse, alcoholism or drug use and are unable to quit or have mental disorders;
* The investigator judges other conditions that may affect the progress of the clinical study and the judgment of the research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Three months
  Complete response rate and partial response rate: measured according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 by means of computed tomography (CT) or magnetic resonance imaging (MRI) at each follow-up.
Adverse events rate | Three months
  Adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Two years
  Defined as the time from randomization until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.
Overall survival (OS) | Two years
  defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chen, M.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China